CLINICAL TRIAL: NCT01334619
Title: Ropivacaine Volume for Ultrasound-guided Retrograde Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Xiaoguang Zhang, Department of Anesthesiology, Beijing Jishuitan Hosptial
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: JSTMZ.2
Record Dates: First submitted 2011-04-07; First posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2010-02

CONDITIONS: Upper Extremity Injury Trauma
Keywords: Anesthetic techniques,regional; Drug delivery,volume; Anesthetic, local: ropivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ropivacaine volume titration (Other)
  Interventions: Procedure: appropriate volume of 0.5% ropivacaine

INTERVENTIONS:
Procedure: appropriate volume of 0.5% ropivacaine — initial concentration: 30 ml, subsequently varied at a ratio of 1: 1.2 for each consecutive patient according to the response of the previous patient, until 5 up-and-down cycles completed.
  Other Names: Naropin

SUMMARY:
The retrograde infraclavicular brachial plexus block has been proved an effective and safe approach. Realtime ultrasound guide will facilitate a successful peripheral nerve block. The purpose of this study was to determine the medium effective volume required to produce an effective retrograde infraclavicular block using an ultrasound (US)-guided technique.

DETAILED DESCRIPTION:
Thirty adults undergoing elective upper limb surgery received an US-guided retrograde infraclavicular block. The initial concentration of 0.5% ropivacaine injected was 30 ml, which was subsequently varied at a ratio of 1: 1.2 for each consecutive patient according to the response of the previous patient. The medium effective volume (EV50) was determined using the Dixon and Massey up-and-down method. The effective volume in 95% of patients (EV95) was calculated using probit regression.

ELIGIBILITY:
Inclusion Criteria:

* Elected upper extremity operations
* BMI 17~30kg/m2
* ASA I/II

Exclusion Criteria:

* Infection at injection site
* Sepsis
* Coagulation Dysfunction
* Phrenic nerve palsy
* Pneumothorax
* Recurrent laryngeal nerve palsy
* Clavicle fracture combined with nerve damage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
VAS of brachial plexus innervated area | 20 minutes
  effect and side effects of the present block approach for brachial plexus.

SECONDARY OUTCOMES:
medium effective ropivacaine volume | about 2 months
  The initial concentration of 0.5% ropivacaine injected was 30 ml, which was subsequently varied at a ratio of 1: 1.2 for each consecutive patient according to the response of the previous patient. The medium effective volume (EV50) was determined using the Dixon and Massey up-and-down method. EV95 was calculated using probit regression.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoguang Zhang, MB, Principal Investigator — Department of Anesthesiology, Beijing Jishuitan Hospital, Beijing, China
Locations (1):
- Beijing jishuitan hospital, Beijing, China